CLINICAL TRIAL: NCT03713372
Title: A Study of Evaluating Recombinant Human Anti-EGFR Monoclonal Antibody (SCT200) for Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma After Failure of Platinum-based Therapy
Brief Title: Safety and Efficacy of SCT200 in Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT200R/MHNSCCII; CTR20181541 (Registry Identifier: China Food and Drug Administration)
Record Dates: First submitted 2018-09-29; First posted 2018-10-19 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Epidermal growth factor receptor; EGFR; SCT200
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-EGFR monoclonal antibody (Experimental): 6.0mg/kg of SCT200 will be administered once a week for a maximum of 6 cycles. After 6 cycles, 8.0mg/kg of SCT200 will be administered every two weeks until disease progression.
  Interventions: Drug: Anti-EGFR monoclonal antibody

INTERVENTIONS:
Drug: Anti-EGFR monoclonal antibody — Initially, 6.0mg/kg of SCT200 will be administered once a week for a maximum of 6 cycles. After 6 cycles, 8.0mg/kg of SCT200 will be administered every two weeks until disease progression.
  Other Names: SCT200

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-EGFR monoclonal antibody（SCT200）in patients with Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma after failure of platinum-based therapy.

DETAILED DESCRIPTION:
This open label, single-arm and multicenter phase II study is designed to evaluate Objective Response Rate (ORR) of anti-EGFR monoclonal antibody（SCT200）in Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma after failure of platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this clinical trial and sign an informed consent form;
* Male or female, age ≥ 18 and ≤ 75 years old;
* The estimated survival period is ≥ 3 months;
* ECOG fitness status score 0 to 1;
* Recurrent and/or metastatic HNSCC (except nasopharyngeal carcinoma) diagnosed by pathology and unable to receive topical treatment (surgery or radiotherapy);
* Patients who have been treated with platinum (cisplatin/carboplatin/nidaplatin) and have clear disease progression during treatment (at least 2 cycles) or after treatment (see RECIST version 1.1) or side effects Intolerance, and the minimum dose of platinum drugs must meet:

  * Minimum dose of cisplatin: ≥60mg/m2 per cycle, or ≥120mg/m2 in 8 weeks;
  * The minimum dose of carboplatin: AUC ≥ 4 / cycle, or total AUC ≥ 8 within 8 weeks.
  * If cisplatin is converted to platinum, the platinum dosage can be calculated using the following formula: carboplatin 1AUC = cisplatin 15mg/m2;
  * The minimum dose of nedaplatin: ≥80mg/m2 per cycle, or ≥160mg/m2 in 8 weeks; Note: Platinum drugs can be used as adjuvant therapy for postoperative patients (synchronous radiotherapy), for palliative chemotherapy in patients with advanced stage or in patients with recurrent and/or metastatic disease.
* Laboratory inspection:

  * Blood routine: neutrophils ≥1.5×l09/L, platelets≥75×109/L, hemoglobin≥80g/L;
  * Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ALT and AST ≤ upper limit of normal value × 3 for liver metastasis, ALT and AST ≤ upper limit of normal value for liver metastases × 5; total bilirubin ( TBIL) ≤ upper limit of normal value × 1.5;
  * Renal function: creatinine (Cr) ≤ normal upper limit × 1.5;
  * Electrolyte: Magnesium ≥ normal lower limit;
* According to the RECIST standard version 1.1, there is at least one measurable tumor lesion. For lesions that have received previous radiotherapy, the target lesion can only be selected if there is a clear disease progression 3 months after the end of radiotherapy.

Exclusion Criteria:

* Patients with a history of central nervous system metastasis or a history of central nervous system metastasis before screening. For patients with clinically suspected central nervous system metastasis, imaging confirmation must be performed within 28 days prior to enrollment to exclude central nervous system metastasis;
* There are other medical history of malignant tumors, except that the malignant lesions have been treated with therapeutic measures 5 years or more before enrollment and there are no known active lesions. The investigator judges that the risk of recurrence is low; Non-melanoma skin cancer, and no evidence of worsening disease; adequately treated cervical cancer in situ, and no evidence of worsening disease; prostatic intraepithelial neoplasia, no evidence of prostate cancer recurrence;
* known to be allergic to antibodies or other components contained in the test drug;
* have received EGFR antibodies (such as panitumumab, cetuximab or its analogs), or small molecule EGFR inhibitors (such as gefitinib, erlotinib, lapatinib, etc.);
* In the 4 weeks or 4 weeks before enrollment, they received anti-tumor drugs (such as chemotherapy, hormone therapy, immunotherapy, antibody therapy, radiotherapy, etc.) or received research drug treatment and could not be included in the evaluation by the investigator. Pain-free palliative radiotherapy for bones;
* At the time of enrollment, patients still had ≥2 toxic side effects (except for hair loss, hearing loss, tinnitus, dry mouth or platinum-induced grade 2 neurotoxicity) caused by previous anti-tumor treatment;
* Patients have been enrolled in other study devices or study drug studies at screening time, or have been deactivated for less than or equal to 4 weeks from other study drugs or study devices;
* Conduct or plan major surgery within 4 weeks prior to enrollment;
* Received transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 2 weeks prior to enrollment;
* Clinically significant cardiovascular disease (defined as: unstable angina, symptomatic congestive heart failure (New York Heart Association [NYHA] ≥ II), uncontrollable severe arrhythmia);
* Myocardial infarction occurred within 6 months prior to enrollment;
* History of interstitial lung disease (ILD), such as interstitial pneumonia, pulmonary fibrosis, or evidence of ILD on baseline chest CT or MRI;
* have clinical symptoms, require clinical intervention or serous effusion (such as pleural effusion and ascites) with a stabilization time of less than 4 weeks;
* medical or psychiatric history or laboratory abnormal medical history that may interfere with the interpretation of the results;
* Patients who are pregnant or breast-feeding, or who plan to be pregnant during the treatment period and within 6 months after the end of treatment;
* Patients (including male or female patients) who are unwilling to receive effective contraception during the treatment period and within 6 months after the end of treatment;
* HCV antibody positive; or HIV positive; or HBV test results: HBsAg positive and / or HBcAb positive and HBV DNA ≥ 104 copy number or ≥ 2000 IU / ml;
* Patients have active or uncontrollable infections (except for simple urinary tract infections or upper respiratory tract infections) requiring systemic treatment within 2 weeks or 2 weeks prior to enrollment;
* known patients have alcohol or drug addiction;
* The investigator believes that patients have other conditions that may affect their adherence to protocol adherence and study indicators, and are not suitable for patients participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-05-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1 year
  The achievement of any stable disease（SD）, partial response (PR) or complete response (CR), according to RECIST v1.1 criteria.
Progresssion free survival(PFS) | 1 year
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 criteria.
Overall survival(OS) | 1 year
  OS is defined as time from first dose of SCT200 until the date of death from any cause.
Immunogenicity | 1 year
  Serum anti-SCT200 antibody levels before and after administration
EORTC QLQ-C30 | 1 year
  Median scores for each item and domain will be reported at each time point. 30 items questionnaire with answers ranging from 1=not at all to 4=very much includes five functional scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, nausea & vomiting and pain) and a global health status/QOL scale. Furthermore, it contains six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties)
EORTC QLQ-H&N35 | 1 year
  European organization for research and treatment of cancer quality of life questionnaire head and neck 35(EORTC QLQ-H & N 35) is a specific questionnaire developed by the European Organisation for Research and Treatment of Cancer for head and neck cancer. The module includes 35 questions Assessing symptoms and side effects of treatment, social function and body image/sexuality .This scale includes seven symptoms subscales that measure pain, swallowing, senses problems, speech problems, trouble with social eating, trouble with social Contact, and less sexuality, and also has 11 subscales related with teeth, opening mouth, dry mouth, sticky saliva, coughing, ill feeling, weight loss, weight gain, use of painkillers, nutritional supplements, and feeding tubes. Standardize the original scores, with scores ranging from 0 to 100, with higher scores representing more serious problems.

CONTACTS AND LOCATIONS:
Overall Officials: yuankai shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No